CLINICAL TRIAL: NCT00396214
Title: A Randomized, Multicenter, Double-Blind, Parallel Group Study To Compare the Effects of Bifeprunox and Quetiapine on Weight Changes in Stable Schizophrenic Patients
Brief Title: Compare the Effects of Bifeprunox and Quetiapine on Weight Changes in Stable Schizophrenic Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This trial discontinued on 2 May 2008 due to lack of enrolment
Sponsor: Solvay Pharmaceuticals (Industry)
Collaborators: H. Lundbeck A/S (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Loretta Stallings, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S154.3.021; 2006-004973-83
Record Dates: First submitted 2006-11-03; First posted 2006-11-06 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; weight changes
MeSH Terms: conditions — Schizophrenia; Body Weight Changes | interventions — bifeprunox; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Bifeprunox
- 2 (Experimental)
  Interventions: Drug: Bifeprunox
- 3 (Active Comparator)
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Bifeprunox — 52 weeks of fixed oral doses of bifeprunox at 30 mg/day administered as a single dose with 1 week upward titration from 0.25 mg/day dose. Placebo will be used for evening dose.
  Arms: 1
Drug: Quetiapine — Fixed oral dose of quetiapine at 400 mg/day to be administered in divided doses (BID) utilizing a 5-day upward titration from 50 mg/day.
  Arms: 3
Drug: Bifeprunox — 52 weeks of fixed oral doses of bifeprunox at 30 mg/day administered as a single dose with 2 week upward titration from 0.25 mg/day dose. Placebo will be used for evening dose.
  Arms: 2

SUMMARY:
The primary objective of the study is to evaluate changes in weight short and long term with bifeprunox and quetiapine. Study participation for the subject is 57 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia
* 18-65 years
* No hospitalization for an exacerbation of schizophrenia within two months prior to screening and during the screening period

Exclusion Criteria:

* Subjects who are acutely psychotic or subjects with current Axis I primary psychiatric diagnosis other than schizophrenia
* At significant risk of suicide, and the potential for violent behavior (likely to harm themselves or others) based on history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Weight | 8 weeks

SECONDARY OUTCOMES:
Change from baseline in Triglyceride | 8 weeks
Detorioration (composite definition using PANSS total score and CGI-I) | 26 weeks
Change from baseline in Weight, Triglyceride and Cardiovascular risk factors | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (151):
- United States (69):
  - Site 313, Anaheim, California
  - Site 333, Anaheim, California
  - Site 323, Cerritos, California
  - Site 374, Costa Mesa, California
  - Site 326, Culver City, California
  - Site 300, Glendale, California
  - Site 343, Long Beach, California
  - Site 356, Los Angeles, California
  - Site 367, Los Angeles, California
  - Site 322, Oceanside, California
  - Site 316, Pasadena, California
  - Site 302, Sacramento, California
  - Site 315, San Diego, California
  - Site 331, San Diego, California
  - Site 340, San Diego, California
  - Site 311, Santa Ana, California
  - Site 336, Santa Ana, California
  - Site 344, Torrance, California
  - Site 318, Denver, Colorado
  - Site 371, Darien, Connecticut
  - Site 358, Hartford, Connecticut
  - Site 360, New Britain, Connecticut
  - Site 317, Hialeah, Florida
  - Site 362, Largo, Florida
  - Site 327, Miami, Florida
  - Site 373, Miami, Florida
  - Site 334, North Miami, Florida
  - Site 351, North Miami, Florida
  - Site 338, Orange City, Florida
  - Site 332, Tampa, Florida
  - Site 330, Atlanta, Georgia
  - Site 308, Augusta, Georgia
  - Site 370, Decatur, Georgia
  - Site 366, Smyma, Georgia
  - Site 337, Chicago, Illinois
  - Site 361, Oakbrook Terrace, Illinois
  - Site 335, Indianapolis, Indiana
  - Site 341, Lake Charles, Louisiana
  - Site 304, Shreveport, Louisiana
  - Site 301, Glen Burnie, Maryland
  - Site 342, Towson, Maryland
  - Site 328, Detroit, Michigan
  - Site 357, Minneapolis, Minnesota
  - Site 309, St Louis, Missouri
  - Site 369, Omaha, Nebraska
  - Site 320, Clementon, New Jersey
  - Site 347, Clementon, New Jersey
  - Site 310, Buffalo, New York
  - Site 312, Buffalo, New York
  - Site 306, Cedarhurst, New York
  - Site 321, New York, New York
  - Site 353, New York, New York
  - Site 372, New York, New York
  - Site 324, Staten Island, New York
  - Site 329, Cincinnati, Ohio
  - Site 345, Oklahoma City, Oklahoma
  - Site 368, Oklahoma City, Oklahoma
  - Site 354, Portland, Oregon
  - Site 314, Philadelphia, Pennsylvania
  - Site 346, Philadelphia, Pennsylvania
  - Site 348, Philadelphia, Pennsylvania
  - Site 350, Sioux Falls, South Dakota
  - Site 352, Memphis, Tennessee
  - Site 307, Austin, Texas
  - Site 303, Conroe, Texas
  - Site 305, Houston, Texas
  - Site 325, San Antonio, Texas
  - Site 319, Richmond, Virginia
  - Site 349, Spokane, Washington
- Argentina (10):
  - Site 502, Buenos Aires
  - Site 506, Buenos Aires
  - Site 505, Córdoba
  - Site 507, Córdoba
  - Site 508, La Plata
  - Site 355, Little Rock
  - Site 501, Mendoza
  - Site 504, Mendoza
  - Site 509, Mendoza
  - Site 503, Rosario
- Canada (12):
  - Site 406, Kelowna, British Columbia
  - Site 411, Victoria, British Columbia
  - Site 408, Halifax, Nova Scotia
  - Site 400, Burlington, Ontario
  - Site 401, Chatham, Ontario
  - Site 404, Mississauga, Ontario
  - Site 407, Orléans, Ontario
  - Site 405, Ottawa, Ontario
  - Site 409, Hull, Quebec
  - Site 403, Prince Albert, Saskatchewan
  - Site 410, Saskatoon, Saskatchewan
  - Site 413, Sydney
- Chile (10):
  - Site 514, Coquimbo
  - Site 510, Santiago
  - Site 511, Santiago
  - Site 512, Santiago
  - Site 513, Santiago
  - Site 516, Santiago
  - Site 517, Santiago
  - Site 518, Santiago
  - Site 519, Santiago
  - Site 515, Valdivia
- Czechia (7):
  - Site 636, České Budějovice
  - Site 637, Kutná Hora
  - Site 604, Litoměřice
  - Site 600, Olomouc
  - Site 601, Pilsen
  - Site 602, Prague
  - Site 605, Prague
- Estonia (3):
  - Site 606, Tallinn
  - Site 608, Tartu
  - Site 607, Võru
- Finland (3):
  - Site 609, Helsinki
  - Site 611, Helsinki
  - Site 610, Turku
- Germany (8):
  - Site 612, Berlin
  - Site 613, Berlin
  - Site 617, Berlin
  - Site 620, Berlin
  - Site 619, Bochum-Gerthe
  - Site 616, Bonn
  - Site 615, München
  - Site 618, Siegen
- Hungary (5):
  - Site 621, Balassagyarmat
  - Site 623, Budapest
  - Site 624, Győr
  - Site 625, Gyula
  - Site 622, Pécs
- Latvia (3):
  - Site 627, Jelgava
  - Site 628, Kaunas
  - Site 626, Sigulda
- Lithuania (2):
  - Site 630, Šilutė
  - Site 629, Vilnius
- Peru (6):
  - Site 520, Lima
  - Site 521, Lima
  - Site 522, Lima
  - Site 523, Lima
  - Site 524, Lima
  - Site 525, Lima
- Slovakia (5):
  - Site 631, Bojnice
  - Site 634, Bratislava
  - Site 632, Liptovský Mikuláš
  - Site 635, Michalovce
  - Site 633, Rimavská Sobota
- South Africa (8):
  - Site 707, Aucklandpark
  - Site 703, Bellair
  - Site 700, Cape Town
  - Site 705, Cape Town
  - Site 706, Cape Town
  - Site 702, Johannesburg
  - Site 701, Pretoria
  - Site 704, Pretoria